CLINICAL TRIAL: NCT04339894
Title: Prospective Epidemiological Study Evaluating the Prevalence of Upper Limb Venous Thrombosis in a Population of Patients Hospitalized in a University Hospital
Brief Title: Prospective Epidemiological Study of Upper Limb Venous Thrombosis
Acronym: Epi-TVMS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0121
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Venous Thrombosis
Keywords: Upper limb; Venous thrombosis; Prevalence; Epidemiology
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Duplex ultrasonography (data collection by extra-corporeal non-invasive sensors) — Search for venous thrombosis and description of thrombosis

SUMMARY:
Venous thrombosis of the upper limb is one of the manifestations of venous thromboembolic disease.

The epidemiology and management of upper limb venous thrombosis is much less well documented than that of lower limb venous thrombosis.

The investigators wished to provide epidemiological data concerning upper limb venous thrombosis in the hospital setting.

The researchers would like to know the prevalence of this pathology among patients hospitalized in a university hospital center. In order to obtain this prevalence, the investigators wish to carry out a monocentric cross-sectional descriptive study.

DETAILED DESCRIPTION:
Venous thrombosis of the upper limb is one of the manifestations of venous thromboembolic disease.

The epidemiology and management of upper limb venous thrombosis is much less well documented than that of lower limb venous thrombosis.

The investigators wished to provide epidemiological data concerning upper limb venous thrombosis in the hospital setting.

The researchers would like to know the prevalence of this pathology among patients hospitalized in a university hospital center. In order to obtain this prevalence, the investigators wish to carry out a monocentric cross-sectional descriptive study.

The main objective of the study is to define the prevalence of upper limb venous thrombosis in patients hospitalized at Nantes University Hospital.

The secondary objectives are to describe the epidemiology according to the patient's hospitalization sector or the endovenous medical devices used. Another secondary objective is to describe the clinical signs associated with thromboses and their characteristics.

The investigators wish to include major patients hospitalized at the Nantes University Hospital in different sectors (medical, surgical, intensive care units). After collecting the patient's non-opposition, reseachers will carry out a venous duplex ultrasonography of the upper limbs.

Data concerning the hospitalization unit, the patient's comorbidities, the presence of venous tracts or other endo-venous devices, clinical signs and duplex ultrasonography data will be collected using a standardized collection grid.

ELIGIBILITY:
Inclusion Criteria :

* Patient (major, pregnant woman) hospitalized in a department of the Nantes University Hospital and accepting participation in this research

Exclusion Criteria :

* Opposition to the completion of the review, minors, adults under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All major patient hospitalized in a department of the Nantes University Hospital and accepting participation in this research
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of upper limb venous thrombosis | through study completion, an average of 1 year
  Number of upper limb venous thrombosis diagnosed in duplex ultrasonography compared to the number of patients examined.

SECONDARY OUTCOMES:
Epidemiology and description of upper limb venous thrombosis | through study completion, an average of 1 year
  Epidemiology of upper limb venous thrombosis according to the patient's hospitalization sector, the patient's history or the medical devices used (pacemaker, peripheral or central venous line, ...). Description of the clinical signs associated with upper limb venous thrombosis. These clinical signs will be correlated with the echodoppler characteristics of the upper limb venous thrombosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France